CLINICAL TRIAL: NCT05974566
Title: Efficacy and Safety of Finerenone in Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: Efficacy and Safety of Finerenone in Heart Failure With Reduced Ejection Fraction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Director, Chongqing Medical University
Other Study IDs: 2023-07
Record Dates: First submitted 2023-07-16; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Diabetes Mellitus; Diabetic Nephropathies
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFrEF patients who accept finerenone therapy: Patients with HFrEF receive finerenone 10mg or 20mg daily treatment for 3 months in addition to other medications.
- HFrEF patients who accept Spironolactone or eplerenone therapy: Patients with HFrEF receive spironolactone or eplerenone treatment daily treatment for 3 months in addition to other medications.

SUMMARY:
Finerenone is a new selective nonsteroidal mineral corticoid receptor antagonist (MRA), nowadays it's widely used in type 2 diabetes (T2DM) patients with chronic kidney disease (CKD), the newest trial shows finerenone improve the cardiovascular outcomes among patients with T2DM and CKD especially reduce the risk of hospitalization for heart failure. In patients with diabetic nephropathy, finerenone resulted in lower risks of CKD progression and cardiovascular events. Finerenone shows great potential therapeutic effect in chronic heart failure (CHF) patients with or without T2DM and CKD compared to eplerenone, but there is still no real world study on finerenone in patients with heart failure with reduced ejection fraction (HFrEF) and it's unclear about the effect of finerenone in CHF patients without T2DM and CKD. The investigators will conduct a study to demonstrate the efficacy and safety of finerenone in HFrEF patients compared to other MRAs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* New York Heart Association(NYHA) functional classification II - IV
* LVEF measured by the echocardiogram ≤ 45%
* eGFR>25mL/min/1.73m²

Exclusion Criteria:

* LVEF measured by the echocardiogram > 45%
* History of allergic or hypersensitivity to drugs involved in the trial.
* Patients with a known history of cancer, angioedema, significant congenital heart disease or rheumatic heart disease.
* Patients diagnosed with myocarditis.
* Probable alternative diagnoses could account for the patient's HF symptoms e.g., COPD, bronchial asthma, primary pulmonary hypertension.
* Systolic blood pressure (SBP) ≥180mmHg or diastolic blood pressure (DBP)

  * 120mmHg at visit, DBP≤90mmHg or symptomatic hypotension.
* Patients with cardiac pacemaker
* Pregnant woman
* eGFR≤25mL/min/1.73m² and not accept long-term hemodialysis therapy.
* Serum potassium >5.2 mmol/l at visit
* Fatal or uncontrollable heart arrythmia e.g., symptomatic or persistence ventricular tachycardia, ventricular rate>150 bpm in AF patients.
* Obvious stenosis (≥50%) of bilateral renal arteries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with heart failure with reduced ejection fraction and NYHA classes II-IV with or without diabetic nephropathy will be incorporated in the study, and other patients who are unable to tolerant treatment will be excluded
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum N-terminal pro-B-type natriuretic peptide (NT-proBNP) | before and after 6 months of medication
  The change in serum NT-proBNP levels in patients was measured before medication and after 6 months of medication to determine the improvement on heart failure

SECONDARY OUTCOMES:
Composite endpoint of death and heart failure rehospitalization | during the 6-month period of medication therapy
  The composite endpoint include the death due to cardiovascular reasons, worsening of renal disease, rehospitalization due to heart failure and admission to hospital to accept intravenous diuretics therapy
Change in left ventricular ejection fraction (LVEF) | before and after 6 months of medication
  The change in LVEF measured by echocardiogram
Change in extracellular volume (ECV) | Before and after 3 months of continuous treatment
  Extracellular volume (ECV) measured by cardiac magnetic resonance imaging (CMR) helps to demonstrate the improvement in myocardial fibrosis
Change in renal function level | Before and after 3 months of continuous treatment
  Change in estimated glomerular filtration rate(eGFR) reflect the renal function

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, PhD, Study Chair — First Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pitt B, Filippatos G, Agarwal R, Anker SD, Bakris GL, Rossing P, Joseph A, Kolkhof P, Nowack C, Schloemer P, Ruilope LM; FIGARO-DKD Investigators. Cardiovascular Events with Finerenone in Kidney Disease and Type 2 Diabetes. N Engl J Med. 2021 Dec 9;385(24):2252-2263. doi: 10.1056/NEJMoa2110956. Epub 2021 Aug 28. PMID 34449181
- [Result] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Nowack C, Schloemer P, Joseph A, Filippatos G; FIDELIO-DKD Investigators. Effect of Finerenone on Chronic Kidney Disease Outcomes in Type 2 Diabetes. N Engl J Med. 2020 Dec 3;383(23):2219-2229. doi: 10.1056/NEJMoa2025845. Epub 2020 Oct 23. PMID 33264825
- [Result] Filippatos G, Anker SD, Bohm M, Gheorghiade M, Kober L, Krum H, Maggioni AP, Ponikowski P, Voors AA, Zannad F, Kim SY, Nowack C, Palombo G, Kolkhof P, Kimmeskamp-Kirschbaum N, Pieper A, Pitt B. A randomized controlled study of finerenone vs. eplerenone in patients with worsening chronic heart failure and diabetes mellitus and/or chronic kidney disease. Eur Heart J. 2016 Jul 14;37(27):2105-14. doi: 10.1093/eurheartj/ehw132. Epub 2016 Apr 29. PMID 27130705